CLINICAL TRIAL: NCT00359801
Title: An International, Multicenter, Large Simple Trial To Evaluate The Long-Term Pulmonary And Cardiovascular Safety Of Exubera In Patients With Diabetes Mellitus
Brief Title: Exubera Large Simple Trial To Evaluate Long-Term Pulmonary And Cardiovascular Safety
Acronym: VOLUME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171069
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus
Keywords: Large Simple Trial
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exubera (Experimental)
  Interventions: Drug: Randomization to Exubera (insulin human [rDNA origin] inhalation powder) or Usual Diabetes Care
- Usual Diabetes Care (Active Comparator)
  Interventions: Drug: Randomization to Exubera (insulin human [rDNA origin] inhalation powder) or Usual Diabetes Care

INTERVENTIONS:
Drug: Randomization to Exubera (insulin human [rDNA origin] inhalation powder) or Usual Diabetes Care — Subjects are randomized to use Exubera. Following initial use of randomized treatment, physicians and subjects are free to change regimens and dosing based on subject response to assigned treatment (as consistent with routine practice). Enrolling physicians are provided with the approved local label for Exubera to guide prescribing and treatment decisions.
  Arms: Exubera
Drug: Randomization to Exubera (insulin human [rDNA origin] inhalation powder) or Usual Diabetes Care — Subjects are randomized to use usual diabetes care. Following initial use of randomized treatment, physicians and subjects are free to change regimens and dosing based on subject response to assigned treatment (as consistent with routine practice).
  Other Names: Non-Exubera
  Arms: Usual Diabetes Care

SUMMARY:
The purpose of this study is to evaluate the long-term pulmonary and cardiovascular safety of Exubera in routine clinical practice.

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera. At that time, Pfizer committed to continued marketing until it returned the licensing rights for the technology to Nektar. Following the announcement, enrollment was halted. Subjects already enrolled and receiving treatment at the time of the halt in enrollment could continue in the study in accordance with the protocol. Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera. As a result, an amendment was filed on April 16, 2008 specifying that all subjects randomized to Exubera had to be transitioned to usual diabetes care, and all study subjects followed for serious adverse events for 6 months. In accordance with this amendment, study A2171069 was terminated on April 29, 2009. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for receiving Exubera treatment based on the approved local label

Exclusion Criteria:

* Pregnant or lactating
* Have a progressive fatal disease or a life expectancy that prohibits them from participating in a five-year research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1976 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (183):
- United States (124):
  - Pfizer Investigational Site, Bay Minette, Alabama
  - Pfizer Investigational Site, Fairhope, Alabama
  - Pfizer Investigational Site, Graysville, Alabama
  - Pfizer Investigational Site, Pell City, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Forrest City, Arkansas
  - Pfizer Investigational Site, Searcy, Arkansas
  - Pfizer Investigational Site, Cudahy, California
  - Pfizer Investigational Site, El Cajon, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Rolling Hills Estates, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Westminster, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Milford, Connecticut
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, DeBary, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Green Cove Springs, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Marianna, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Niceville, Florida
  - Pfizer Investigational Site, Opa-locka, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Warner Robins, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Greenville, Illinois
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Bossier City, Louisiana
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Elkton, Maryland
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Plymouth, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Battle Creek, Michigan
  - Pfizer Investigational Site, Clinton, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Muskegon, Michigan
  - Pfizer Investigational Site, Sterling Heights, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Warren, Michigan
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Grand Island, Nebraska
  - Pfizer Investigational Site, Incline Village, Nevada
  - Pfizer Investigational Site, Belleville, New Jersey
  - Pfizer Investigational Site, Belvidere, New Jersey
  - Pfizer Investigational Site, Glendora, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Babylon, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New Hartford, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Asheboro, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Morehead City, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Shelby, North Carolina
  - Pfizer Investigational Site, Tabor City, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bismarck, North Dakota
  - Pfizer Investigational Site, Ashtabula, Ohio
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, McConnelsville, Ohio
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Clinton, Oklahoma
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Broomall, Pennsylvania
  - Pfizer Investigational Site, Dauphin, Pennsylvania
  - Pfizer Investigational Site, Fogelsville, Pennsylvania
  - Pfizer Investigational Site, Hanover, Pennsylvania
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Jeannette, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Jersey Shore, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Plymouth Meeting, Pennsylvania
  - Pfizer Investigational Site, Tipton, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Florence, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, North Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Garland, Texas
  - Pfizer Investigational Site, Hurst, Texas
  - Pfizer Investigational Site, Kaufman, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Stephenville, Texas
  - Pfizer Investigational Site, Webster, Texas
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Ettrick, Virginia
  - Pfizer Investigational Site, Burnsville, West Virginia
  - Pfizer Investigational Site, Charleston, West Virginia
- Germany (40):
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Doberan
  - Pfizer Investigational Site, Bad Grönenbach
  - Pfizer Investigational Site, Bad Oeynhausen
  - Pfizer Investigational Site, Bad Staffelstein
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Datteln
  - Pfizer Investigational Site, Dortmund
  - Pfizer Investigational Site, Eisenach
  - Pfizer Investigational Site, Emden
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Esslingen am Neckar
  - Pfizer Investigational Site, Falkensee
  - Pfizer Investigational Site, Friedberg
  - Pfizer Investigational Site, Fulda
  - Pfizer Investigational Site, Hagen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hohenmölsen
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Leverkusen
  - Pfizer Investigational Site, Mahlberg
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, Markdorf
  - Pfizer Investigational Site, Marl
  - Pfizer Investigational Site, Meissen
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Neuwied
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Reinfeld
  - Pfizer Investigational Site, Riesa
  - Pfizer Investigational Site, Schlüchtern
  - Pfizer Investigational Site, Siegen
  - Pfizer Investigational Site, Suhl
  - Pfizer Investigational Site, Villingen-Schwenningen
  - Pfizer Investigational Site, Wangen
  - Pfizer Investigational Site, Wangen I. Allgaeu
  - Pfizer Investigational Site, Warburg
- Pfizer Investigational Site, Manatí, Puerto Rico
- Sweden (4):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Forshaga
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lilla Edet
- United Kingdom (14):
  - Pfizer Investigational Site, Chesterfield, Derbyshire
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Dronfield, Sheffield
  - Pfizer Investigational Site, Weybridge, SURREY
  - Pfizer Investigational Site, Woking, Surrey
  - Pfizer Investigational Site, Rugby, Warwickshire
  - Pfizer Investigational Site, Warminster, WILTSHIRE
  - Pfizer Investigational Site, Sheffield, Yorkshire
  - Pfizer Investigational Site, Airdrie
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Westbury

REFERENCES:
- [Derived] Gatto NM, Bracken MB, Kolitsopoulos F, Duggan WT, Koch GG, Wise RA, Jackson NC. Pulmonary and cardiovascular safety of inhaled insulin in routine practice: The Exubera Large Simple Trial (VOLUME). Contemp Clin Trials Commun. 2019 Aug 13;18:100427. doi: 10.1016/j.conctc.2019.100427. eCollection 2020 Jun. PMID 32478195
- [Derived] Kolitsopoulos FM, Gatto NM, Sweetland K, Bracken MB, Jackson N. Implications of product withdrawal on a post-approval pragmatic trial: The VOLUME study experience. Contemp Clin Trials Commun. 2019 Oct 28;16:100477. doi: 10.1016/j.conctc.2019.100477. eCollection 2019 Dec. PMID 31799472
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171069&StudyName=Exubera%20Large%20Simple%20Trial%20To%20Evaluate%20Long-Term%20Pulmonary%20And%20Cardiovascular%20Safety

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from primary care centers, diabetes and endocrinology clinics, and academic centers, and participated in the study between 22 July 2006 and 29 April 2009.
Groups:
- Exubera®: Exubera® plus usual diabetes care
- Non-Exubera®: Usual diabetes care
Period: Overall Study
Arm/Group | Exubera® | Non-Exubera®
Started | 987 | 989
Completed | 682 (7 additional subjects had missing data and final status (completed/discontinued) is unknown.) | 769 (4 additional subjects had missing data and final status (completed/discontinued) is unknown.)
Not Completed | 305 | 220
Not completed — Lost to Follow-up | 72 | 58
Not completed — Withdrawal by Subject | 143 | 96
Not completed — Other | 66 | 46
Not completed — Final Status Unknown: missing data | 7 | 4
Not completed — Sponsor Decision | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exubera® | Non-Exubera® | Total
Number analyzed (Participants) | 987 | 989 | 1976
Age, Customized [Number; unit: participants]
  18-44 years | 114 | 133 | 247
  45-64 years | 576 | 552 | 1128
  65-74 years | 242 | 245 | 487
  75-84 years | 52 | 57 | 109
  >= 85 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 439 | 434 | 873
  Male | 548 | 555 | 1103

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Decline in Forced Expiratory Volume (FEV1) Exceeding 20% From Baseline
Description: Persistent decline in FEV1 exceeding 20% from baseline: observed decline in FEV1 exceeding 20% from baseline, 3 months after a confirmed decline (2 consecutive declines within 1 month) in FEV1 exceeding 20% from baseline. Second pulmonary function test (PFT) that confirmed decline was to occur within 14-42 days of the decline. Persistence: PFT that established persistence was to occur within 60-120 days of the confirming (2nd) decline. Index Visit: date subject had final Scheduled spirometry; was to occur within 2 months of Institutional Review Board/Ethics approval of April 2008 amendment.
Time Frame: Baseline, Month 6, Year 1, Year 2, Index Visit
Population: Full Analysis Set: all randomized subjects.
Measure: Number; unit: participants
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
participants
  Initial FEV1 Decline | 100 | 112
  Initial FEV1 Decline but not a Confirmed Decline | 81 | 105
  Confirmed FEV1 Decline | 19 | 7
  Confirmed FEV1 Decline but not Persistent Decline | 11 | 7
  Persistent FEV1 Decline | 8 | 0

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: Change from Baseline: mean of value of observed forced expiratory volume in the first second of forced exhalation [FEV1] in liters [L] at observation minus Baseline value. Index Visit: date subject had final scheduled spirometry; was to occur within 2 months of Institutional Review Board/Ethics approval of April 2008 amendment.
Time Frame: Baseline, Week 26, Week 52, Week 104, Index Visit
Population: FAS; (n) = number of subjects with analyzable data at observation for Exubera® and Non-Exubera®, respectively.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
liters
  Baseline (n=985, 987) | 2.661 (0.838) | 2.684 (0.888)
  Week 26 (n=813, 852) | -0.009 (0.568) | -0.035 (0.509)
  Week 52 (n=470, 482) | -0.032 (0.411) | -0.056 (0.465)
  Week 104 (n=3, 1) | -0.103 (0.607) | -1.270 (0.000)
  Index Visit (n=729, 803) | -0.000 (0.559) | -0.018 (0.580)

3. Secondary Outcome: Pulmonary Serious Adverse Event (SAE) Composite: SAEs of Asthma, Chronic Obstructive Pulmonary Disease (COPD), Pneumonia, or Acute Bronchitis
Description: Endpoint committee adjudicated the endpoint based on review of medical and hospital records, and results were classified using standard criteria. Definite: definite pneumonia, definite COPD, or definite asthma; possible: possible pneumonia, possible COPD, possible asthma, probable obstructive lung disease not otherwise specified or probable acute bronchitis; definite or possible: either definite or possible; insufficient: insufficient data.
Time Frame: Baseline through End of Study
Population: FAS
Measure: Number; unit: events
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
events
  Definite | 4 | 1
  Possible | 3 | 2
  Definite or Possible | 7 | 3
  Insufficient | 4 | 2

4. Secondary Outcome: Time to Event for Pulmonary Serious Adverse Event (SAE) Composite: SAEs of Asthma, Chronic Obstructive Pulmonary Disease (COPD), Pneumonia, or Acute Bronchitis
Description: Elapsed time, in days, from the start of a subject's participation in the study to the date of the first report of an event subsequently confirmed (according to protocol definition) as meeting the criteria for pulmonary SAE composite. Censoring time: elapsed time, in days, from the start of a subject's participation in the study to the latest contact with the subject for the particular analysis set of interest. Cox proportional hazards model to estimate treatment effect.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, originally planned inferential analysis for time to event was not done.
Measure: Number; unit: days
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: All-cause Mortality: Number of Deaths
Description: Endpoint committee adjudicated the endpoint based on review of medical and hospital records, and results were classified using standard criteria (confirmation of deaths by blinded adjudicator(s) through medical records or death certificates). Patients meeting the endpoint All Cause Mortality after adjudication by the endpoint committee.
Time Frame: Baseline through End of Study
Population: FAS
Measure: Number; unit: participants
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
participants | 12 | 9

6. Secondary Outcome: Time to Event: All-cause Mortality
Description: Time to all-cause mortality: elapsed time, in days, from the start of a subject's participation in the study to the date of the event subsequently confirmed (according to protocol definition) as meeting the criteria for all-cause mortality. Censoring time: elapsed time, in days, from the start of a subject's participation in the study to the latest contact with the subject for the particular analysis set of interest. Cox proportional hazards model to estimate treatment effect.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, originally planned inferential analysis for time to event was not done.
Measure: Number; unit: days
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Supplemental Definition of Decline in Forced Expiratory Volume in One Second (FEV1): Number of Subjects
Description: Confirmed FEV1 decline: any two consecutive declines that are >= 14 days apart. The pulmonary function test that established persistence occured >= 60 days after the initial decline. A confirmed decline: any two consecutive declines ≥ 14 days apart. The third PFT that established persistence was to occur ≥ 60 days after the initial decline. Index Visit: date the subject had his/her final scheduled spirometry was to occur within 2 months of Institutional Review Board/Ethics approval of April 2008 amendment.
Time Frame: Baseline, Month 6, Year 1, Year 2, Index Visit
Population: FAS
Measure: Number; unit: participants
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
participants
  Initial FEV1 Decline | 100 | 112
  Initial FEV1 Decline but not a Confirmed Decline | 62 | 74
  Confirmed FEV1 Decline | 38 | 38
  Confirmed FEV1 Decline but not Persistent Decline | 11 | 14
  Persistent FEV1 Decline | 27 | 24

8. Secondary Outcome: Cardiovascular SAE Composite: SAEs of Cardiovascular Mortality, Non-fatal Myocardial Infarction (MI), or Non-fatal Stroke
Description: Endpoint committee adjudicated based on review of medical/hospital records; results classified using standard criteria. Definite: definite MI or stroke; Possible: possible MI or stroke; Other (non-MI, non-stroke): other cardiovascular event (non-MI, non-stroke); Definite or possible: either definite or possible or both; Insufficient: insufficient data; Death from cardiovascular or cerebrovascular: cardiovascular or cerebrovascular event; Definite or possible or death from cardiovascular or cerebrovascular: either definite or possible or both or cardiovascular or cerebrovascular event.
Time Frame: Baseline through End of Study
Population: FAS
Measure: Number; unit: events
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
events
  Definite | 5 | 3
  Possible | 5 | 6
  Other (non-myocardial infarction, non-stroke) | 15 | 9
  Definite or Possible | 10 | 9
  Insufficient | 9 | 7
  Death from Cardiovascular or Cerebrovascular | 2 | 4
  Definite or Possible, or Death from Cardiovascular | 12 | 11

9. Secondary Outcome: Time to Event for Cardiovascular Serious Adverse Event (SAE) Composite: SAEs of Cardiovascular Mortality, Non-fatal Myocardial Infarction, or Non-fatal Stroke
Description: Elapsed time, in days, from the start of a subject's participation in the study to the date of the first event subsequently confirmed (according to protocol definition) as meeting the criteria for cardiovascular SAE composite. Censoring time: elapsed time, in days, from the start of a subject's participation in the study to the latest contact with the subject for the particular analysis set of interest. Cox proportional hazards model to estimate treatment effect.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, originally planned inferential analysis for time to event was not done.
Measure: Number; unit: days
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Allergic Response Serious Adverse Event (SAE) Composite: SAEs of Anaphylaxis, Angioedema, Generalized Allergic Reaction, or Allergic Bronchospasm
Description: Endpoint committee adjudicated the endpoint based on review of medical and hospital records, and results were classified using standard criteria. Definite or possible: anaphylaxis, angioedema/urticaria, bronchospasm or possible allergic reaction not otherwise specified (NOS); Insufficient: insufficient data.
Time Frame: Baseline through End of Study
Population: FAS
Measure: Number; unit: events
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
events
  Definite or Possible | 2 | 0
  Insufficient | 3 | 0

11. Secondary Outcome: Time to Event for Allergic Response Serious Adverse Event (SAE) Composite, Including: SAEs of Anaphylaxis, Angioedema, Generalized Allergic Reaction, or Allergic Bronchospasm
Description: Elapsed time, in days, from the start of a subject's participation in the study to the date of the first event subsequently confirmed (according to protocol definition) as meeting the criteria for allergic response. Censoring time: elapsed time, in days, from the start of a subject's participation in the study to the latest contact with the subject for the particular analysis set of interest. Cox proportional hazards model to estimate treatment effect.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, originally planned inferential analysis for time to event was not done.
Measure: Number; unit: days
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline
Description: Baseline HbA1c: the latest determination prior to beginning study participation. Change from Baseline: HbA1c at observation (falling within the time window associated with a given analysis set) minus the baseline value.
Time Frame: Baseline, Month 6, Year 1, Year 2, Index Visit
Population: FAS; (n) = number of subjects with analyzable data at observation for Exubera® and Non-Exubera®, respectively.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 987 | 989
percent
  Baseline (n=978, 985) | 8.6 (1.9) | 8.5 (1.9)
  Week 26: Observed Value (804, 849) | 8.0 (1.8) | 8.0 (1.8)
  Week 26: Change from Baseline (n=800, 848) | -0.5 (1.7) | -0.5 (1.6)
  Week 52: Observed Value (n=468, 489) | 7.8 (1.7) | 7.7 (1.6)
  Week 52: Change from Baseline (n=467, 489) | -0.4 (1.6) | -0.6 (1.6)
  Week 104: Observed Value (n=3, 1) | 6.6 (1.2) | 6.0 (0)
  Week 104: Change from Baseline (n=3, 1) | -1.0 (1.6) | -2.7 (0)
  Index Visit: Observed Value (n=673, 754) | 8.1 (3.0) | 8.0 (3.5)
  Index Visit: Change from Baseline (n=669, 754) | -0.3 (2.9) | -0.5 (3.3)

13. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline
Description: Baseline HbA1c taken as the latest determination prior to beginning study participation. Change = on-study value (for measurements falling within the time window associated with a given analysis set) minus the baseline value. Linear model with terms for treatment, baseline HbA1c, time on study, and subject within treatment.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, the originally planned inferential analysis (linear model) for change from baseline was not done.
Measure: Number; unit: percent
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Time to Persistent Decline in FEV1 Exceeding 20% From Baseline
Description: Elapsed time, in days, from the start of subject's participation in the study to the first reading of FEV1 that is: 20% or more below the subject's latest pre-study measurement, subsequently confirmed as a >20% decline [(baseline observed value minus visit observed value)/by baseline observed value *100], and assessed as persistent as defined by protocol process. Censoring time: elapsed time, in days, from the start of a subject's participation in the study to latest valid FEV1 measurement for the particular analysis set of interest. Cox proportional hazards model to estimate treatment effect.
Time Frame: Baseline to 5 years
Population: FAS. Due to early study termination, originally planned inferential analysis for time to event was not done.
Measure: Number; unit: days
Arm/Group | Exubera® | Non-Exubera®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Two additional subjects experienced SAEs that were not listed under a treatment group due to data error: Injury, Poisoning and Procedural Complications system organ class (1 subject; drug exposure during preganancy), and Musculoskeletal and Connective System Disorders System Organ Class (1 subject; neuropathic arthropathy).
Arm/Group | Exubera® | Non-Exubera®
Serious Adverse Events (participants affected / at risk) | 124/987 | 109/989
Other Adverse Events (participants affected / at risk) | 26/987 | 11/989
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exubera® (N=987) | Non-Exubera® (N=989)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphatic obstruction (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 2 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Cerebral palsy (Congenital, familial and genetic disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Eye degenerative disorder (Eye disorders) | 0 | 1
Macular oedema (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 7 | 9
Death (General disorders) | 2 | 1
Discomfort (General disorders) | 1 | 0
Drug ineffective (General disorders) | 2 | 0
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Organ failure (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Device occlusion (Injury, poisoning and procedural complications) | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Paternal drugs affecting foetus (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Anti-insulin antibody increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 3 | 0
Catheterisation cardiac (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 6
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 3
Convulsion (Nervous system disorders) | 0 | 4
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 4
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Hydroureter (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac operation (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 1
Toe amputation (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exubera® (N=987) | Non-Exubera® (N=989)
Angina pectoris (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 3 | 0
Cardiac murmur (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Stent placement (Surgical and medical procedures) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Pursuant to Pfizer's announcement that it would exit marketing of Exubera®, study enrollment was halted on 26-October-2007.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.